CLINICAL TRIAL: NCT01300455
Title: A Study to Evaluate the Effects of MK-4305 in Patients With Obstructive Sleep Apnea
Brief Title: Effects of Suvorexant in Participants With Obstructive Sleep Apnea (MK-4305-036)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4305-036
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Sleep Apnea
Keywords: Insomnia; obstructive sleep apnea; orexin receptor antagonist
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders; Sleep Apnea, Obstructive | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suvorexant (40 mg) (Experimental): In Period 1, suvorexant (40 mg tablets) administered orally once daily for 4 consecutive days in the evening. Period 1 is followed by a washout period of a minimum of 5 days. Period 2 consists of placebo administered once daily for 4 consecutive days in the evening.
  Interventions: Drug: Suvorexant; Drug: Matching Placebo
- Placebo (Placebo Comparator): In Period 1, placebo administered orally once daily for 4 consecutive days in the evening. Period 1 is followed by a washout period of a minimum of 5 days. In Period 2, suvorexant (40 mg tablets) administered once daily for 4 consecutive days in the evening.
  Interventions: Drug: Suvorexant; Drug: Matching Placebo

INTERVENTIONS:
Drug: Suvorexant — 40 mg tablets, orally once daily for 4 consecutive days in the evening
  Other Names: MK-4305; SCH 900433
Drug: Matching Placebo — Placebo tablets, orally once daily for 4 consecutive days in the evening

SUMMARY:
This study will evaluate the safety, tolerability, and effect of multiple doses of suvorexant (MK-4305) on respiratory function in participants with mild to moderate obstructive sleep apnea (OSA) compared to administration of placebo. The primary hypothesis of this study is that multiple doses of MK-4305 do not produce a clinically significant increase in Apnea-Hypopnea Index (AHI) in participants with mild to moderate OSA, as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of reproductive potential must demonstrate a serum β-human chorionic gonadotrophin (hCG) level consistent with the nongravid state at the pre-study (screening) visit and agree to use (and/or have their partner use) two (2) acceptable methods of birth control beginning at the pre-study visit throughout the study.
* Women who are postmenopausal without menses for at least 1 year and a follicle stimulating hormone (FSH) value in the postmenopausal range upon pre-study (screening) evaluation, and/or are status post hysterectomy, oophorectomy or tubal ligation may participate.
* Participants with a Body Mass Index (BMI) ≤40 kg/m2 at the pre-study (screening) visit.
* Participants have to be in good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests.
* Participants without clinically significant abnormality on electrocardiogram (ECG) performed at the pre-study (screening) visit and/or prior to administration of the initial dose of study drug.
* Participants have an International Classification of Sleep Disorders diagnosis of OSA.
* Participants have confirmed mild or moderate OSA (defined as mild

OSA with AHI ≥5 and <15, and moderate OSA with AHI ≥15 and <30) based on the screening nighttime polysomnography (NPSG).

* Participants have a usual bedtime between 20:00 (8:00 post meridiem [PM]) and 00:30 (12:30 ante meridiem [AM)] and is not subject to any other unusual changes in sleeping routine and sleeps for 4 hours or more per night.
* Participants must complete a sleep history diary for at least 5 consecutive days and up to 21 days prior to the screening PSG visit.
* Participant has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months; participants who have discontinued smoking or the use of nicotine/nicotine containing products for at least approximately 3 months may be enrolled in the study at the discretion of the investigator.

Exclusion Criteria:

* Participants have used continuous positive airway pressure devise (CPAP) or a dental appliance within the preceding 7 days prior to screening NPSG Visit, or is required to use CPAP or a dental appliance during course of the study (7 days prior to the screening NPSG, throughout the study [including washout intervals between treatment periods], and until the poststudy visit).
* Participants have other than OSA and evidence of another clinically significant, active pulmonary disorder such as bronchiectasis, emphysema, or asthma documented by history, physical examination, or chest x-ray.
* Participant have either a history within the past 6 months prior to the prestudy visit or current evidence of an unstable or clinically significant cardiovascular disorder, including but not limited to acute coronary syndrome, unstable angina, congestive heart failure, cardiogenic syncope, cardiomyopathy, any symptomatic arrhythmia, orthostatic hypotension, or uncontrolled hypertension.
* Participants have abnormal pre-randomization laboratory values other clinically significant, unexplained laboratory abnormality in the opinion of the investigator with alanine transaminase (ALT) >1.5 x the upper limit of normal (x ULN), aspartate transaminase (AST) >1.5 x ULN, total bilirubin >1.5 x ULN, or serum creatinine of >2 mg/dL.
* Participants have a history or diagnosis of narcolepsy, cataplexy (familial or idiopathic), circadian rhythm sleep disorder, parasomnia including nightmare disorder, sleep terror disorder, sleepwalking disorder, and REM behavior disorder, periodic limb movement (PLM) disorder, restless legs syndrome, or primary hypersomnia.
* Participants have a screening PSG recording with oxygen (O2) saturation <80% for ≥5% of the total sleep time, and >10 PLM per hour associated with an arousal (periodic limb movement arousal index [PLMAI]).
* Participant is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 to 10 years. Participant who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Participant has lifetime history of bipolar disorder, a psychotic disorder, or posttraumatic stress disorder; or, a psychiatric condition requiring treatment with a prohibited medication; or, other psychiatric condition that, in the investigator's opinion, would interfere with the participant's ability to participate in the study.
* Participant, in the opinion of the investigator, has a history or current evidence of any condition, therapy, lab or ECG abnormality or other circumstances that might confound the results of the study, or interfere with the participant's participation for the full duration of the study.
* Participant has any history of a neurological disorder, including but not limited to seizure disorder (other than single episodes of childhood febrile seizures), stroke, transient ischemic attack, multiple sclerosis, cognitive impairment, or significant head trauma with sustained loss of consciousness within the last 10 years.
* Participant has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases. Participants with a history of uncomplicated kidney stones may be enrolled in the study at the discretion of the investigator.
* Participant has a history of neoplastic disease except: 1. adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix may participate in the study; 2. participants with other malignancies which have been successfully treated ≥10 years prior to the prestudy (screening) visit where, in the judgment of both the Investigator and treating physician, appropriate follow-up has revealed no evidence of recurrence from the time of treatment through the time of the prestudy (screening) visit, or 3. participants, who, in the opinion of the Investigator, are highly unlikely to sustain a recurrence for the duration of the study.
* Participant is a nursing mother.
* Participant has a positive screening urine alcohol test or drug test.
* Participant has a need for more than 3 toilet visits during the night.
* Participant is taking, or plans to take, one or more of prohibited concomitant medication.
* Participant consumes excessive amounts of alcohol (greater than 3 glasses of alcoholic beverages), excessive amounts of coffee, tea, cola, or other caffeinated beverages per day.
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy (screening) visit.
* Participant has a history of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
* Participant is currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years.
* Participant works a night shift and is not able to avoid night shift work within 2 weeks before each treatment visit (or before the study start and during the study).
* Participant has traveled across 3 or more time zones (transmeridian travel) in the last 1 week prior to study start.
* Participant is at imminent risk of self-harm or harm to others
* Any concern by the investigator regarding the safe participation of the participant in the study or for any other reason; the investigator considers the participant inappropriate for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03-19 (Actual); Primary Completion 2011-08-11 (Actual); Study Completion 2011-08-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Sun H, Palcza J, Card D, Gipson A, Rosenberg R, Kryger M, Lines C, Wagner JA, Troyer MD. Effects of Suvorexant, an Orexin Receptor Antagonist, on Respiration during Sleep In Patients with Obstructive Sleep Apnea. J Clin Sleep Med. 2016 Jan;12(1):9-17. doi: 10.5664/jcsm.5382. PMID 26194728
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=4305-036&kw=4305-036&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Suvorexant (40 mg) Then Placebo: In Period 1, suvorexant (40 mg tablets) administered orally, once daily, for 4 consecutive days in the evening. Period 1 is followed by a washout period of a minimum of 5 days. Period 2 consists of placebo administered once daily for 4 consecutive days in the evening.
- Placebo Then Suvorexant (40 mg): Period 1 consists of placebo administered once daily for 4 consecutive days in the evening. Period 1 is followed by a washout period of a minimum of 5 days. In Period 2, suvorexant (40 mg tablets) administered orally, once daily, for 4 consecutive days in the evening.
Period: Period 1
Arm/Group | Suvorexant (40 mg) Then Placebo | Placebo Then Suvorexant (40 mg)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Washout
Arm/Group | Suvorexant (40 mg) Then Placebo | Placebo Then Suvorexant (40 mg)
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Suvorexant (40 mg) Then Placebo | Placebo Then Suvorexant (40 mg)
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant (40 mg) Then Placebo | Placebo Then Suvorexant (40 mg) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: years] | 48 [34 to 63] | 50 [30 to 64] | 49 [30 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Apnea-Hypopnea Index (AHI)
Description: Evaluation of the effect of multiple dose administration of suvorexant on
  AHI as measured by polysomnography. The AHI is an overall index of obstructive sleep apnea (OSA) severity. The AHI is calculated by dividing the number of apneas and hypopneas by the number of hours of sleep. AHI values are categorized as mild OSA = 5 to <15/hr and moderate OSA = 15 to <30/hr.
Time Frame: Day 4
Population: Twenty-five of 26 participants had Day 4 data; one participant did not receive placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per hour
Groups:
- Suvorexant (40 mg): Participants administered a 40-mg dose of suvorexant.
- Placebo: Participants administered placebo.
Arm/Group | Suvorexant (40 mg) | Placebo
Number analyzed (Participants) | 26 | 25
Events per hour | 17.07 [13.30 to 20.84] | 14.41 [10.61 to 18.22]
Statistical Analysis 1: Comparison: Suvorexant (40 mg) vs Placebo; Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 2.66, 90% CI 2-sided [0.22 to 5.09]

2. Primary Outcome: Number of Participants With an Adverse Event
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 14 days after last dose
Population: All participants were included in the Safety Population.
Measure: Number; unit: participants
Arm/Group | Suvorexant (40 mg) | Placebo
Number analyzed (Participants) | 26 | 26
participants | 8 | 4

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 13 days
Population: All participants were included in the Safety Population.
Measure: Number; unit: participants
Arm/Group | Suvorexant (40 mg) | Placebo
Number analyzed (Participants) | 26 | 26
participants | 0 | 0

4. Secondary Outcome: Mean Arterial Oxygen Saturation (SaO2) During Total Sleep Time
Description: Evaluation of the effect of multidose dose suvorexant on mean SaO2 during total sleep time as measured by pulse oximetry. Total sleep time is the total of all rapid eye movement (REM) and non-REM sleep in a sleep episode.
Time Frame: Day 1 and Day 4
Population: Twenty-four of 26 participants were included in the primary evaluation of Day 1 AHI/SaO2 data; 2 participants had no data due to either not receiving placebo or an equipment malfunction. Twenty-five of 26 participants had Day 4 data; one participant did not receive placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Oxygen Saturation
Arm/Group | Suvorexant (40 mg) | Placebo
Number analyzed (Participants) | 26 | 25
Percentage of Oxygen Saturation
  Day 1 (n = 26, 24) | 94.12 [93.48 to 94.75] | 94.15 [93.50 to 94.80]
  Day 4 (n = 26, 25) | 94.15 [93.53 to 94.78] | 94.21 [93.59 to 94.84]
Statistical Analysis 1: Comparison: Suvorexant (40 mg) vs Placebo; Day 1, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Mean Difference (Final Values) = -0.04, 90% CI 2-sided [-0.49 to 0.42]
Statistical Analysis 2: Comparison: Suvorexant (40 mg) vs Placebo; Day 4, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = -0.06, 90% CI 2-sided [-0.45 to 0.33]

5. Secondary Outcome: Percentage of Total Sleep Time That Arterial SaO2 is Less Than 90%, 85%, and 80%
Description: Evaluation of the percentage of the night in which SaO2 is less than 90%, less
  than 85% and less than 80% following multiple dose administration of
  suvorexant and placebo. Total sleep time is the total of all REM and non-REM sleep in a sleep episode.
Time Frame: Day 1 and Day 4
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Percentage of Total Sleep Time
Arm/Group | Suvorexant (40 mg) | Placebo
Number analyzed (Participants) | 26 | 25
Percentage of Total Sleep Time
  Day 1 (SaO2 is less than 90%) (n = 26, 24) | 3.31 [1.03 to 5.58] | 2.57 [0.22 to 4.92]
  Day 1 (SaO2 is less than 85%) (n = 26, 24) | 0.48 [0.12 to 0.85] | 0.24 [-0.14 to 0.61]
  Day 1 (SaO2 is less than 80%) (n = 26, 24) | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted. | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted.
  Day 4 (SaO2 is less than 90%) (n = 26, 25) | 2.16 [0.88 to 3.45] | 1.95 [0.66 to 3.25]
  Day 4 (SaO2 is less than 85%) (n = 26, 25) | 0.69 [0.16 to 1.23] | 0.41 [-0.13 to 0.95]
  Day 4 (SaO2 is less than 80%) (n = 26, 25) | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted. | NA [NA to NA] — Due to the small number of participants experiencing SaO2 less than 80%, a formal statistical analysis was not conducted.
Statistical Analysis 1: Comparison: Suvorexant (40 mg) vs Placebo; Day 1, SaO2 <90%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Mean Difference (Final Values) = 0.74, 90% CI 2-sided [-1.31 to 2.79]
Statistical Analysis 2: Comparison: Suvorexant (40 mg) vs Placebo; Day 1, SaO2 <85%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Mean Difference (Final Values) = 0.25, 90% CI 2-sided [-0.10 to 0.59]
Statistical Analysis 3: Comparison: Suvorexant (40 mg) vs Placebo; Day 4, SaO2 <90%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Mean Difference (Final Values) = 0.21, 90% CI 2-sided [-0.59 to 1.01]
Statistical Analysis 4: Comparison: Suvorexant (40 mg) vs Placebo; Day 4, SaO2 <85%, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [-0.09 to 0.65]

6. Secondary Outcome: Mean Arterial SaO2 for Different Sleep Stages
Description: Comparison of the mean SaO2 during different sleep stages (REM, Non-REM, and awake) following multiple dose administration of suvorexant and placebo. Sleep stages were determined by polysomnography.
Time Frame: Day 1 and Day 4
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Oxygen Saturation
Arm/Group | Suvorexant (40 mg) | Placebo
Number analyzed (Participants) | 26 | 25
Percentage of Oxygen Saturation
  Day 1 - Mean SaO2 During REM (n = 26, 24) | 94.08 [93.34 to 94.82] | 94.14 [93.38 to 94.90]
  Day 1 - Mean SaO2 during Non-REM (n = 26, 24) | 94.12 [93.47 to 94.76] | 94.07 [93.41 to 94.73]
  Day 1 - Mean SaO2 during Wake (n = 26, 24) | 94.42 [93.74 to 95.11] | 94.94 [94.23 to 95.65]
  Day 4 - Mean SaO2 During REM (n = 26, 25) | 93.96 [93.17 to 94.76] | 93.83 [93.03 to 94.63]
  Day 4 - Mean SaO2 during Non-REM (n = 26, 25) | 94.27 [93.64 to 94.90] | 94.25 [93.62 to 94.89]
  Day 4 - Mean SaO2 during Wake (n = 26, 25) | 94.73 [94.11 to 95.36] | 94.91 [94.28 to 95.54]
Statistical Analysis 1: Comparison: Suvorexant (40 mg) vs Placebo; Day 1, REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of Least Squares Means; Mean Difference (Final Values) = -0.06, 90% CI 2-sided [-0.61 to 0.49]
Statistical Analysis 2: Comparison: Suvorexant (40 mg) vs Placebo; Day 1, Non-REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Sqares Means; Mean Difference (Final Values) = 0.05, 90% CI 2-sided [-0.41 to 0.50]
Statistical Analysis 3: Comparison: Suvorexant (40 mg) vs Placebo; Day 1, Wake, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = -0.51, 90% CI 2-sided [-1.13 to 0.10]
Statistical Analysis 4: Comparison: Suvorexant (40 mg) vs Placebo; Day 4, REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of the Least Squares Means; Mean Difference (Final Values) = 0.13, 90% CI 2-sided [-0.24 to 0.50]
Statistical Analysis 5: Comparison: Suvorexant (40 mg) vs Placebo; Day 4, Non-REM, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Median Difference (Final Values) = 0.02, 90% CI 2-sided [-0.40 to 0.43]
Statistical Analysis 6: Comparison: Suvorexant (40 mg) vs Placebo; Day 4, Wake, Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference in the Least Squares Means; Median Difference (Final Values) = -0.18, 90% CI 2-sided [-0.61 to 0.25]

7. Secondary Outcome: Mean AHI
Description: Evaluation of the effect of multiple dose administration of suvorexant on
  AHI as measured by polysomnography. The AHI is an overall index of OSA severity. The AHI is calculated by dividing the number of apneas and hypopneas by the number of hours of sleep. AHI values are categorized as mild OSA = 5 to <15/hr and moderate OSA = 15 to <30/hr.
Time Frame: Day 1
Population: Twenty-four of 26 participants were included in the primary evaluation of Day 1 AHI/SaO2 data; 2 participants had no data due to either not receiving placebo or an equipment malfunction.
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per hour
Arm/Group | Suvorexant (40 mg) | Placebo
Number analyzed (Participants) | 26 | 24
Events per hour | 16.25 [12.65 to 19.86] | 16.72 [13.02 to 20.42]
Statistical Analysis 1: Comparison: Suvorexant (40 mg) vs Placebo; Difference (Suvorexant - Placebo) of Least Squares Means; Test type: Superiority or Other; Difference of Least Squares Means; Mean Difference (Final Values) = -0.47, 90% CI 2-sided [-3.20 to 2.26]

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose
Arm/Group | Suvorexant (40 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 5/26 | 2/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant (40 mg) (N=26) | Placebo (N=26)
Nausea (Gastrointestinal disorders) | 0 | 2
Somnolence (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.